CLINICAL TRIAL: NCT00661037
Title: SAFEty of Two Strategies of ICD Management at Implantation
Acronym: SAFE-ICD
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 2007_SI
Record Dates: First submitted 2008-04-07; First posted 2008-04-18 (Estimated); Results first posted 2017-06-20 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-06

CONDITIONS: Ventricular Fibrillation; Ventricular Flutter; Sudden Cardiac Death
MeSH Terms: conditions — Ventricular Fibrillation; Ventricular Flutter; Death, Sudden, Cardiac | interventions — Defibrillators, Implantable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Patients having VF induction with shock termination at implant
  Interventions: Device: Implantable defibrillator
- 2: Patients not having VF induction at implant or during follow-up
  Interventions: Device: Implantable defibrillator

INTERVENTIONS:
Device: Implantable defibrillator — Implantable defibrillator to reduce ventricular arrhythmias via shock.
  Other Names: Not applicable. All devices allowed.
  Groups: 1
Device: Implantable defibrillator — Implantable defibrillator to reduce ventricular arrhythmias via shock.
  Other Names: Not applicable. All devices allowed.
  Groups: 2

SUMMARY:
The aim of this prospective observational study is to evaluate the safety, over a follow-up of 2 years, of two strategies, consisting in performing or not performing defibrillation testing(DT) during first implant of implantable cardioverter defibrillator

DETAILED DESCRIPTION:
The standardized requirements for implantable cardioverter defibrillator (ICD) include defibrillation testing (DT), consisting in induction and termination of ventricular fibrillation (VF). An effective DT has historically been considered part of standard procedures at implant. Nevertheless, implant techniques and technology have evolved during years and nowadays deviations are frequent in clinical practice mainly due to the fact that physicians are seriously concerned about the risk of severe complications related to DT. However, the practice of not performing DT is arbitrary and its safety is yet unproven. This observational study will assess the safety of the two strategies adopted at ICD implant: induction (including patients who undergo DT at implant) and non-induction (including patients who do not undergo DT at implant. No deviation from the centres' current practice in choosing to perform or not perform DT is introduced by this study protocol. The study considers consecutive patients undergoing first implant of ICD

ELIGIBILITY:
Inclusion Criteria:

* first implantation of ICD or CRT-D
* Patients undergoing upgrade to ICD or CRT-D from pacemaker
* Patients undergoing upgrade to CRT-D from CRT
* Age 18 or above, or legal age to give written informed consent

Exclusion Criteria:

* Patients who do not give consent to treat their data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients having the risk of life threatening arrhythmias and indicated for the implant of an implantable cardioverter defibrillator.
Sampling Method: Non-Probability Sample
Enrollment: 2120 (Actual)
Dates: Start 2008-03; Primary Completion 2011-05 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michele Brignole, MD, Study Chair — Ospedali del Tigullio
Locations (1):
- Ospedali del Tigullio, via Don Bobbio 25, Lavagna, Italy

REFERENCES:
- [Derived] Brignole M, Occhetta E, Bongiorni MG, Proclemer A, Favale S, Iacopino S, Calo L, Vado A, Buja G, Mascioli G, Quartieri F, Tritto M, Parravicini U, Castro A, Tomasi C, Villani GQ, D'Acri MG, Klersy C, Gasparini M; SAFE-ICD Study Investigators. Clinical evaluation of defibrillation testing in an unselected population of 2,120 consecutive patients undergoing first implantable cardioverter-defibrillator implant. J Am Coll Cardiol. 2012 Sep 11;60(11):981-7. doi: 10.1016/j.jacc.2012.05.014. Epub 2012 Aug 1. PMID 22858384

RESULTS

PARTICIPANT FLOW:
Groups:
- VF Induction: Patients having VF induction with shock termination at implant (Implantable defibrillator: Implantable defibrillator to reduce ventricular arrhythmias via shock)
- no VF Induction: Patients not having VF induction at implant or during follow-up
  Implantable defibrillator: Implantable defibrillator to reduce ventricular arrhythmias via shock.
Period: Overall Study
Arm/Group | VF Induction | no VF Induction
Started | 836 | 1284
Witdrawn | 47 | 68
Deaths | 108 | 188
Completed | 682 | 1027
Not Completed | 154 | 257

BASELINE CHARACTERISTICS:
Groups:
- no VF Induction: Patients not having VF induction at implant or during follow-up (Implantable defibrillator: Implantable defibrillator to reduce ventricular arrhythmias via shock)
- Total: Total of all reporting groups
Arm/Group | VF Induction | no VF Induction | Total
Number analyzed (Participants) | 836 | 1284 | 2120
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (12) | 67 (11) | 66 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 152 | 268 | 420
  Male | 684 | 1016 | 1700
Region of Enrollment [Number; unit: participants]
  Italy | 836 | 1284 | 2120

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Severe Intra-operative Complications at ICD Implant and/or Events at Follow up
Description: * Severe implant-related* complications at ICD implants among the following:
    * Survival from cardiopulmonary arrest due to VF requiring 3 or more consecutive external shocks for termination or due to electro-mechanical dissociation.
    * Transient ischemic attack or stroke,
    * Cardiogenic shock,
    * Pulmonary edema,
    * Embolic events,
    * Anoxic coma
    * Pericardial tamponade
    * Death.
  * Events at follow up:
    * Sudden cardiac death (defined as witnessed unexpected death occurring <1 hour from symptoms onset or unwitnessed during sleep)
    * Resuscitation after ineffective documented appropriate ICD shocks
      * Implant related events are considered as those listed above, occurring during the implant procedure in the timeframe betweend device poket insertion and patient exit from the cath-lab, as well as those events occurring after the patient exit from the cath-lab that, after review from the event adjudication committee, have been classified as related to the implant procedure.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | VF Induction | no VF Induction
Number analyzed (Participants) | 836 | 1284
Participants | 18 | 16

2. Secondary Outcome: Severe Intra-operative Complications
Description: including: cardiopulmonary arrest, transient ischemic attack or stroke, cardiogenic shock, pulmonary edema, embolic event, anoxic coma, pericardial tamponade,death
Time Frame: Acute (ICD implant)
Measure: Count of Participants; unit: Participants
Arm/Group | VF Induction | no VF Induction
Number analyzed (Participants) | 836 | 1284
Participants | 8 | 4

3. Secondary Outcome: Sudden Cardiac Death at Follow up or Resusciation After Ineffective Documented Appropriate ICD Shocks at Follow up
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Groups:
- VF Induction: Patients having VF induction with shock termination at implant
- No- VF Induction: Patients not having VF induction at implant or during follow-up
Arm/Group | VF Induction | No- VF Induction
Number analyzed (Participants) | 836 | 1284
Participants | 10 | 12

ADVERSE EVENTS:
Time Frame: 2 years
Description: Adverse Events were assessed without regard to the specific Adverse Event Terms but classified withing the boundaries of ISO classfication: Adverse Event (AE); Adverse Device Effect (ADE); Serious Adverse Event (SAE): Serious Adverse Device Effect (SADE)
Arm/Group | VF Induction | no VF Induction
All-Cause Mortality (participants affected / at risk) | 108/836 | 188/1284
Serious Adverse Events (participants affected / at risk) | 209/836 | 177/1284
Other Adverse Events (participants affected / at risk) | 120/836 | 90/1284
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VF Induction (N=836) | no VF Induction (N=1284)
SAE-serious adverse events (Cardiac disorders) | 146 (222) | 133 (205)
SADE - serious adverse device effects (Cardiac disorders) | 63 (107) | 44 (74)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VF Induction (N=836) | no VF Induction (N=1284)
AE - Adverse Events (Non serious / non device related) (Cardiac disorders) | 42 (53) | 44 (53)
ADE - non serious adverse device effects (Cardiac disorders) | 78 (126) | 46 (70)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No